CLINICAL TRIAL: NCT04428840
Title: Effects of Implementation of Automated Pre-triage Based on a Self-measurement Kiosk With Questionnaire for Patients in the Emergency Department Waiting Room on Triage Time-stamps and Satisfaction of Use
Brief Title: Effects of Implementation of a Self-measurement Kiosk in the Emergency Department Waiting Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spoedopname (Other)
Responsible Party: Sponsor-Investigator, Spoedopname, Professor Peter De Paepe, University Hospital, Ghent
Organization: University Hospital, Ghent (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019/0315
Record Dates: First submitted 2019-11-12; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Emergencies
Keywords: triage; kiosk; early warning score
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: Patients are randomised in blocks per day regarding use of the kiosk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- on-day (Experimental): Use of the self-measurement kiosk: measurement of vital signs + completion of short questionnaire
  Interventions: Device: Self-measurement kiosk
- Off-day (No Intervention): No use of the self-measurement kiosk

INTERVENTIONS:
Device: Self-measurement kiosk — Use of the self-measurement kiosk, with results forwarded to the triage nurse screens
  Other Names: BeWell kiosk
  Arms: on-day

SUMMARY:
In this study the participant will be invited to be seated in the self-measurement kiosk after registration in the Emergency department. In this kiosk, the participant will be measuring their own vitals and answering a short questionnaire regarding the reason for presentation. All these results are displayed on a screen for the triage nurse. Based on the results, high-risk patients will be highlighted on the screen, so they may be seen faster.

DETAILED DESCRIPTION:
The questionnaire entails questions which would otherwise be asked by the triage nurse, regarding reason for presentation, fever, pain and and possible allergies. This is done through a touch-screen.

The vital signs and potential alarm symptoms from the (multilingual) questionnaire are being displayed with the pain score on a screen in the triage room and at the nurses desk. An adapted Early Warning Score (aEWS - without respiratory rate) is calculated from the vital signs. Abnormal results are being highlighted and carried up on the screen to the top position. This enables the triage nurse to pick up the sicker participants in the waiting room faster. The measurements are valid, so they do not have to be repeated by the triage nurse.

Users will be contacted afterwards regarding satisfaction of use

ELIGIBILITY:
Inclusion Criteria:

* all patients presenting ambulatory at the Emergency Department

Exclusion Criteria:

* patients presenting by ambulance / Emergency Medical Services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 757 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Triage time-stamp 1 | through study completion, average of 1 year
  Shorter time to end of triage process: Time from registration to time of end of triage process (completion of electronic record)
Triage time-stamp 2 | through study completion, average of 1 year
  Shorter time to beginning of triage process: Time from registration to time of start of triage process (initiation of electronic record)

SECONDARY OUTCOMES:
Time to see physician | through study completion, average 1 year
  Shorter time to see physician: Time from registration to start of medical assessment (first of record of physician care)

CONTACTS AND LOCATIONS:
Overall Officials: Cathelijne Lyphout, MSc, Principal Investigator — UZ Gent
Locations (1):
- Spoedgevallendienst, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No
No plan to share - General Data Protection Regulation related